CLINICAL TRIAL: NCT03598127
Title: Vitamin A Status in Critically Ill Children With Sepsis and Its Association With Illness Severity
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Yi Ji, Doctor, West China Hospital
Other Study IDs: 2018-333
Record Dates: First submitted 2018-06-24; First posted 2018-07-26 (Actual); Last update posted 2021-04-08 (Actual); Status verified 2021-04

CONDITIONS: Sepsis
Keywords: Vitamin A; status; sepsis; illness severity
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples are collected from the patients in the first 24h of admission, then the blood samples are centrifuged at 3000 rpm for 5 min to separate the serum.The serum was aliquoted in marked Eppendorf test tubes and frozen at -70℃.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- sepsis group: patients of sepsis group are diagnosed with sepsis according to International Pediatric Sepsis Consensus Conference:Definitions for sepsis and organ dysfunction in pediatrics.
- control group: A gender- and age- matched control group are recruited from among non-sepsis children from Pediatric Intensive Care Unit of West China Hospital.

SUMMARY:
The primary purpose of this study is to assess the status of vitamin A in critically ill children with sepsis and its association with the ill severity. The second purpose is to evaluate the performance of three tools in predicting mortality in our population which are used for measuring the illness severity in pediatric intensive care units.

DETAILED DESCRIPTION:
Sepsis is a worldwide health problem, resulting in million of deaths each year. Sepsis caused by infectious diseases is also a common cause of death in children, and infectious diseases account for more than 50% of the deaths. The prevalence of sepsis and severe sepsis in children steadily rose in past decade. Although tremendous resources and efforts were consumed for the disease, the mechanism of sepsis is still unknown. However, sepsis 3.0 recommended that sepsis should be defined as life-threatening organ dysfunction caused by a dysregulated host response to infection. Study found that sepsis is characterized by a hyperinflammatory immune response in early phase and suppression of immune system in the later phase of sepsis. There are 10% of the deaths in the early phase due to overwhelming inflammation presenting with fever, shock, and multiorgan failure, while 30% of deaths caused by superinfection occur in the later phase.

Vitamin A, one of lipid soluble vitamins, plays an important role in immune system. Vitamin A deficiency increases the risk of infection, and vitamin A deficiency is highly prevalent among children, especially in developing country. Vitamin A is essential for T cells differentiation, induced regulatory T cells (iTregs) and Th17 cells balance, and orchestrating immune responses, etc, which contribute to the immune response in patients with sepsis.Our previous studies revealed that vitamin A deficiency presented in children with enterovirus 71 (EV71) infection was associated with reduced immunity and more severe illness.So we hypothesize that vitamin A or vitamin A deficiency may play an essential role in sepsis. However, data on status of vitamin A or prevalence of vitamin A deficiency in children with sepsis is limited.We conduct a study to to assess the status of vitamin A in critically ill children with sepsis and its association with the illness severity.

There are three widely used score systems for measuring the illness severity in pediatric intensive care units: the pediatric risk of mortality (PRISM), the pediatric index of mortality (PIM) and the pediatric logistic organ dysfunction (PELOD) score. Though the three systems are validated in other populations, they are not commonly used in our population because lack of validation. We will evaluate the performance of the three tools in our population simultaneously in this study.

ELIGIBILITY:
Inclusion Criteria:

* Age ≤16 years old
* Diagnose of sepsis
* Consent of both parents (or the person having parental authority in families)

Exclusion Criteria:

* Discharging against medical advise
* Age>16 years
* Condition of underlying chronic disease (hepatic, renal, cardiac,neurological, pulmonary and gastrointestinal)
* Patients with haematological malignancies and immunodeficiency

(As for evaluating the performance of the three score systems, all patients admitted to the PICU are included except adolescents >16 years of age and those patients who stayed in the PICU for < 2h.)

Ages: 0 Months to 192 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Patients admitted to the pediatric intensive care unit of West China Hospital of Sichuan University are screened and recruited.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2018-06-01 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Comparison of vitamin A levels between sepsis group and control group,and assessment of VA status in sepsis patients with and without organ dysfunction | 1 year
  Demographic data(age in months, gender, race, weight in kilograms) are collected. VA concentrations of the serum samples measured by mg/dl are analyzed by high-performance liquid chromatography. Laboratory test results (serum creatinine in mmol/L, total bilirubin in mg/dL, PaCO2 in mmHg, and platelet count per mm^3, etc) are collected to identify organ dysfunctions.

SECONDARY OUTCOMES:
the association between serum vitamin A concentrations and illness severity in children with sepsis | 1 year
  Severity of illness are measured by Pediatric Risk of Mortality (PRISM) scores, and to investigate the correlation between PRISM scores and A concentrations.
Performance of PRISM in predicting mortality in pediatric intensive care units in Chinese population. | 1 year
  The PRISM scores are accrued from most abnormal values of 14 physiology variables in the first 24h of admission. The minimum score is 0, and maximum is 76 which is almost invariably associated with death.
Performance of PIM2 in predicting mortality | 1 year
  The index of PIM2 are calculate with 10 variables in the fist 1h of admission, and the index is transferred to probability of death.
Performance of PELOD-2 in predicting mortality | 1 year
  The PELOD-2 score include 10 variables, each variable is ranging from 0 to 6 (some are less than 6). the maximum score is 33 and the minimum is 0. Larger the score means worsen status of a patient.

CONTACTS AND LOCATIONS:
Locations (1):
- West China Hospital of Sichuan University, Chengdu, Sichuan, China

REFERENCES:
- [Derived] Zhang X, Sun K, Lu G, Feng L, Chen S, Ji Y. Comparison of PICU Cost and Severity-Adjusted Cost Between Patients With SIRS-Defined Sepsis and Those With Age-Adapted SOFA-Defined Sepsis. Front Pediatr. 2021 Feb 25;9:628918. doi: 10.3389/fped.2021.628918. eCollection 2021. PMID 33718302
- [Derived] Zhang X, Yang K, Chen L, Liao X, Deng L, Chen S, Ji Y. Vitamin A deficiency in critically ill children with sepsis. Crit Care. 2019 Aug 1;23(1):267. doi: 10.1186/s13054-019-2548-9. PMID 31370866